CLINICAL TRIAL: NCT02499185
Title: A PILOT Study Evaluating Novel Biomarkers of AKI in Post-operative Patients Undergoing Major Intra-Abdominal Surgery
Brief Title: Study Evaluating Novel Biomarkers of AKI (Acute Kidney Injury) in Post-operative Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients with renal failure
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NOVELBIO
Record Dates: First submitted 2015-06-30; First posted 2015-07-16 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2016-10

CONDITIONS: Acute Kidney Injury; Arterial Hypertension; Obesity; Cardio Vascular Disease; Diabetes Mellitus; Chronic Liver Disease; Hypercholesterolemia
Keywords: Biomarker; Intra Abdominal Surgery; AKI
MeSH Terms: conditions — Acute Kidney Injury; Hypertension; Obesity; Diabetes Mellitus; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nephro Check Test (Experimental): We take urine samples and analyse the level of [TIMP-2]●[IGFBP-7] using the NephroCheck Test to diagnose AKI
  Interventions: Device: Nephro Check Test; Other: serum creatinine measurement
- serum creatinine measurement (Active Comparator): This is the "Golden standard" to diagnose AKI
  Interventions: Device: Nephro Check Test; Other: serum creatinine measurement

INTERVENTIONS:
Device: Nephro Check Test — Urine sample
Other: serum creatinine measurement — Blood sample

SUMMARY:
To validate the use of [TIMP-2]●[IGFBP-7] to predict AKI in patients undergoing major intra abdominal surgery.

DETAILED DESCRIPTION:
A prospective pilot single center study to investigate the potential of [TIMP-2].[IGFBP-7] to predict AKI (Acute Kidney Injury) in patients undergoing major abdominal surgery. The investigators will measure the biomarker once preoperatively and 4-times postoperatively starting at arrival on PACU (post anesthesia care unit).The primary endpoint of this study is the development of AKI stage 2 or 3 within the first 72 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* High risk patients: General Surgery AKI Risk Index Class III, IV or V
* Major abdominal surgery

Exclusion Criteria:

* Ongoing acute kidney injury Stage 2/3
* History of kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with AKI stage 2 or 3 using the updated rifle "KDIGO" guidelines | 72 Hours

SECONDARY OUTCOMES:
Number of participants who need renal replacement therapy | 30 Days
  the need renal replacement therapy wil be evaluated by the nephrologist (acid base disturbances, hypervolemia,...)

OTHER OUTCOMES:
30-day mortality | 30 days
persistence of renal dysfunction at 30 days | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lien Torisaen, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Jan Poelaert, Prof.Dr., Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No